CLINICAL TRIAL: NCT04880200
Title: The GAIN (Greater Access and Impact With NAT) Study: Improving HIV Diagnosis, Linkage to Care, and Prevention Services With HIV Point-of-Care Nucleic Acid Tests (NATs)
Brief Title: Improving HIV Diagnosis, Linkage to Care, and Prevention Services With HIV Point-of-Care Nucleic Acid Tests
Acronym: GAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joanne Stekler, MD MPH, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00010387; 6 U01 PS 005196-01-01 (Other Grant/Funding Number: CDC); 6U01PS005196 (NIH)
Record Dates: First submitted 2021-04-27; First posted 2021-05-10 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: HIV Infections
Keywords: HIV; point of care testing; nucleic acid testing
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: For the aim #3 RCT, we will randomize participants 1:1 to the POC NAT intervention arm and to standard of care. The intervention will include a SAMBA test and adherence counseling intervention developed by the study team to accompany delivery of test results. The study team will train participating primary care providers (PCPs) in delivery of the adherence counseling intervention.
  Study staff will discuss the study, obtain informed consent, and, for participants randomized to POC NAT, perform SAMBA and provide results to the PCP. Study staff will perform venipuncture, ensure that individual laboratory NAT is performed, and administer a brief CASI. PCPs will deliver the POC NAT result and adherence counseling intervention to patients during their visit. Participants will be asked to sign an ROI that allows the study to share POC NAT results with the PCP and allows the study staff to obtain outcomes measures from clinical patient data for longitudinal follow up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- POC NAT & Adherence Intervention (Experimental): These participants will receive the POC NAT test during their study visit. The result will be conveyed to their provider, who will deliver the result and an adherence intervention.
  Interventions: Diagnostic Test: POC NAT & Adherence Intervention
- Standard of Care (No Intervention): These participants will receive the clinical standard of care during their visit.

INTERVENTIONS:
Diagnostic Test: POC NAT & Adherence Intervention — The POC NAT test will be the SAMBA Semi-Q HIV test. The adherence intervention will be developed by study staff and tailored for delivery along with the POC NAT results.
  Arms: POC NAT & Adherence Intervention

SUMMARY:
This project will develop, implement, and evaluate models for use of point-of-care nucleic acid testing (POC NAT) among HIV-negative persons seeking HIV testing, PEP, and PrEP and HIV-positive persons in community and clinical settings. Study aims #1 and #2 will evaluate the sensitivity and specificity of a qualitative POC NAT in persons not known to be HIV-positive and will determine the impact of its use on PrEP uptake and persistence among persons testing HIV-negative and on time to HIV continuum of care outcomes among persons testing HIV-positive. Aim #3 will implement a POC NAT-tailored behavioral intervention to evaluate impact on time to virologic suppression among PLWH receiving ART. Aim #4 will quantify the acceptability and feasibility of implementation of POC NAT in community and clinical settings and collect cost and related data for cost-effectiveness analyses. Finally, in Aim #5, a distinct but related study will compare the sensitivity, specificity, and agreement of multiple POC NATs over a range of HIV RNA levels.

ELIGIBILITY:
Inclusion Criteria:

* Persons who are HIV-positive and seeking care at Madison Clinic.
* 18 years of age or older
* Patient's provider is willing to deliver adherence intervention
* Patient is getting a laboratory RNA viral load test that day.
* Able to read and speak English

Exclusion Criteria:

* Patients of unknown HIV status
* Patients who have participated in the study before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 932 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Time to viral suppression | Participants will be enrolled for up to 6 months
  We will compare time to virologic suppression among participants randomized to the two arms.

SECONDARY OUTCOMES:
Participation | Participants will be enrolled for up to 6 months
  We will use descriptive statistics to report on the proportion of Madison primary care providers (PCP)s willing to participate in the RCT and the proportion of patients who agree to study enrollment.

OTHER OUTCOMES:
POC NAT limit of detection | Participants will be enrolled for up to 6 months
  We will report on the limit of detection of the SAMBA test, using the plasma HIV RNA level as gold standard, and the agreement (kappa) of SAMBA and plasma HIV RNA level, dichotomized at 1000 copies/mL

CONTACTS AND LOCATIONS:
Overall Officials: Joanne D Stekler, MD, Principal Investigator — University of Washington
Locations (1):
- Madison Clinic, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Intellectual property and data generated will be administered in accordance with UW and CDC policies. Final determinations for data sharing will be based on guidelines for use determined by the Publication Committee. Data obtained during this project will be available at the end of the funding cycle or within a year of publication of major findings, whichever is later. Requests for data or specimens must be made in writing, and human subjects approval must be obtained prior to data transfer. Data will be provided from the Data Center electronically, stripped of identifying information. Investigators receiving data will be asked to sign an agreement stipulating that they will (1) use data only for not-for-profit research purposes (unless negotiated otherwise with the Publication Committee); (2) not attempt to identify any individual participant; (3) secure data using appropriate technology and not share data with anyone else; and (4) destroy data after analyses are completed.